CLINICAL TRIAL: NCT01951521
Title: RandomizEd Controlled Trial for Pre-operAtive Dose-escaLation BOOST in Locally Advanced Rectal Cancer
Brief Title: RECTAL BOOST Study
Acronym: RECTAL BOOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Maastro Clinic, The Netherlands (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Principle Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL46051.041.13
Record Dates: First submitted 2013-09-18; First posted 2013-09-26 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Locally advanced rectal cancer; Radiotherapy; Boost; Dose-escalation; Pathological complete response; Response
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: cohort multiple randomized controlled trial
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Boost (Experimental): Boost radiation consists of 5 fractions of 3 Gy (total 15 Gy) delivered to the tumor (Gross Tumor Volume) additional to standard chemoradiation of 50 Gy with Capecitabine.
  Interventions: Radiation: Boost
- Standard chemoradiation (No Intervention): Standard chemoradiation consisting of 25 x 2 Gy (total 50 Gy) with Capecitabine.

INTERVENTIONS:
Radiation: Boost — External Beam radiation delivered using intensity modulation radiation therapy (IMRT) planning, consisting of 15 Gy (in 5 sequential fractions).
  Arms: Boost

SUMMARY:
Randomized controlled trial in which the effect is investigated of a radiation boost in addition to standard chemoradiation in patients with locally advanced rectal cancer on complete response rate defined as pathological complete response, in those who undergo surgery, or 2-years local recurrence-free survival (2y-LRFS), in those who opted for a wait and see approach. Secondary objectives are adverse events due to chemoradiation (acute, perioperative and late toxicity), tumor response assessed with MRI, the impact of the boost on local and distant recurrence and survival as well as patient-reported quality of life and workability. The need for this comprehensive study is emphasized by the sub-optimal (radiation-) methods, heterogeneity between and poor reporting in the few previous trials in this field.

DETAILED DESCRIPTION:
Rationale: The current treatment for locally advanced rectal cancer consists of pre-operative chemoradiation treatment (CRT) (50 Gray (Gy) in 25 fractions) followed by surgical resection, according to T-/N-stage, circumferential resection margin (CRM) and tumor localization (see table 1). After this neo-adjuvant treatment approximately 15% of patients show pathological complete response (pCR), i.e.no residual tumor in the resected specimen on pathologic examination. Patients with pCR have a lower risk of local and distant recurrences and significantly longer disease-free and overall survival. Furthermore, in these patients surgery could possibly have been omitted. Selected patients with a clinical complete response (cCR), defined prior to surgery by rectoscopy, rectal examination and magnetic resonance imaging (MRI), may opt for an organ-preserving therapy, a so called wait and see approach.

Response to chemoradiation occurs in a dose dependent fashion. Therefore, recent trials aimed to improve prognosis by radiation dose-escalation that resulted in improved pCR rates. Toxicity rates associated with radiation doses above 60 Gy are manageable and differ between studies; from increased to comparable or even lower toxicity. Moreover, dose escalation may increase the proportion of patients eligible for organ-preserving therapy.

Objective: We study whether addition of a radiation boost to standard chemoradiation in patients with locally advanced rectal cancer increases the complete response rate defined as pathological complete response, in those who undergo surgery, or 2-years local recurrence-free survival (2y-LRFS), in those who opted for a wait and see approach. Secondary objectives are adverse events due to chemoradiation (acute, perioperative and late toxicity), tumor response assessed with MRI, the impact of the boost on local and distant recurrence and survival as well as patient-reported quality of life and workability. The need for this comprehensive study is emphasized by the sub-optimal (radiation-) methods, heterogeneity between and poor reporting in the few previous trials in this field.

Study design: Multicentre Randomized Controlled Trial, nested within a prospective cohort according to the 'cohort multiple randomized controlled trial' (cmRCT) design.

Study population: Rectal cancer patients participating in a prospective cohort (the PLCRC project) and diagnosed with adenocarcinoma of the rectum whom will undergo chemoradiation based on clinical criteria (see table 1 section 1.2.1).

Intervention: An irradiation boost of 15 Gy delivered to the gross tumor volume (GTV) in 5 fractions in addition to the standard chemoradiation treatment of 50 Gy. Thereby increasing the total GTV dose to 65 Gy.

Main study parameters/endpoints: The primary endpoint is complete response either defined as pathological complete response (pCR) in patients who undergo surgery, assessed by standardized pathologic examination of the surgical specimen, or 2-years local recurrence-free survival (LRFS) after chemoradiation in patients who opted for a wait and see approach. Secondary outcomes are treatment acute, perioperative and late toxicity, tumor response assessed with MRI, patient-reported quality of life and workability, local recurrence and (disease-specific) survival.

ELIGIBILITY:
Inclusion criteria

* Participant in the PLCRC project (ClinicalTrials.gov: NCT02070146)
* Informed consent obtained for being offered experimental interventions within the PLCRC project
* Informed consent obtained for questionnaires on patient reported outcomes within the PLCRC project
* WHO: 0-2
* Indication for chemoradiation based on primary tumor, regional nodes, metastasis (TNM) stage
* Referred for chemoradiation
* No contra-indication for MRI
* Tumor distance from ano-rectal transition ≤10 cm

Exclusion criteria

* <18 years
* No indication for chemoradiation according to Dutch guidelines based on TNM staging.
* Inflammatory bowel disease
* Prior pelvic radiotherapy
* At least one contra-indication for Capecitabine administration (based on Dihydropyrimidine dehydrogenase (DPD)-deficiency, bloodcount, liver malfunction, renal failure (Creatinine clearance <30 ml/min), medical history such as recent cardiac events
* Recent pregnancy ≤ 1 year ago
* Inadequate understanding of the Dutch language in speech and/or writing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | pathologic examination following surgery, at aproximately 13-15 weeks (control arm) or 14-16 weeks (boost arm) after randomization or clinical complete respons of 2 years after first response assessment.
  The primary endpoint is complete response either defined as pathological complete response (pCR) in patients who undergo surgery, assessed by standardized pathologic examination of the surgical specimen, or 2-years local recurrence-free survival (LRFS) after chemoradiation in patients who opted for a wait and see approach.

SECONDARY OUTCOMES:
Acute toxicity in common toxicity criteria for adverse events (CTCAE). | Until surgery at 8-10 weeks post chemoradiation (which is 13-15 weeks (control) or 14-16 weeks (boost) post randomization
  Outcomes are assessed according to Common Toxicity Criteria for Adverse Events (CTCAE) (v4.0).
Patient reported quality of life | at baseline and 3, 6, 12 and 24 months after treatment.
  at baseline and 3, 6, 12 and 24 months after treatment. Patient reported outcome (Quality of life (QoL)) is measured by validated questionnaires.
  QoL: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and CR-29 (these acronyms indicate cancer and colorectal cancer specific questionnaires.
Tumor response on Magnetic resonance imaging (MRI) | at week 2 during chemoradiation and week 7 post chemoradiation.
  During (week 2) and after (7-8 weeks post) chemoradiation tumor response is assessed by (several) MRI (sequences such as T1, T2 and DWI).
Patient reported workability | at baseline and 3, 6, 12 and 24 months after treatment.
  validated questionnaires. Patient reported outcome (workability) is measured by Workability index.
Surgical complication | untill 30 days after surgery, which is 17-19 weeks (control) or 18-20 weeks (boost) post randomization
  Dutch Surgical Colorectal Audit criteria for surgical complication. This includes wound-infection, wound-healing (time), hospitalization (time), supportive treatment.
(disease-free) survival | up to death of included patients, for a maximum of 60 years post-randomization.
  Survival is measured, as well as other clinical data, in the PICNIC Cohort (ProspectIve data CollectioN Initiative on Colorectal cancer) reviewed by Dutch Medical Ethics Committee @ University Medical Center Utrecht, under number 12-510.

CONTACTS AND LOCATIONS:
Overall Officials: HM Verkooijen, MD PhD, Principal Investigator — Imaging Division, UMC Utrecht; M. Berbee, MD PhD, Principal Investigator — Radiation-Oncology, MAASTRO clinic
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Verweij ME, Hoendervangers S, Couwenberg AM, Burbach JPM, Berbee M, Buijsen J, Roodhart J, Reerink O, Pronk A, Consten ECJ, Smits AB, Heikens JT, van Grevenstein WHMU, Intven MPW, Verkooijen HLM. Impact of Dose-Escalated Chemoradiation on Quality of Life in Patients With Locally Advanced Rectal Cancer: 2-Year Follow-Up of the Randomized RECTAL-BOOST Trial. Int J Radiat Oncol Biol Phys. 2022 Mar 1;112(3):694-703. doi: 10.1016/j.ijrobp.2021.09.052. Epub 2021 Oct 8. PMID 34634436
- [Derived] Couwenberg AM, Burbach JPM, Berbee M, Lacle MM, Arensman R, Raicu MG, Wessels FJ, Verdult J, Roodhart J, Reerink O, Hoendervangers S, Buijsen J, Grabsch HI, Pronk A, Consten ECJ, Smits AB, Heikens JT, Appelt AL, van Grevenstein WMU, Verkooijen HM, Intven MPW. Efficacy of Dose-Escalated Chemoradiation on Complete Tumor Response in Patients with Locally Advanced Rectal Cancer (RECTAL-BOOST): A Phase 2 Randomized Controlled Trial. Int J Radiat Oncol Biol Phys. 2020 Nov 15;108(4):1008-1018. doi: 10.1016/j.ijrobp.2020.06.013. Epub 2020 Jun 19. PMID 32565319
- [Derived] Couwenberg AM, Burbach JPM, May AM, Berbee M, Intven MPW, Verkooijen HM. The trials within cohorts design facilitated efficient patient enrollment and generalizability in oncology setting. J Clin Epidemiol. 2020 Apr;120:33-39. doi: 10.1016/j.jclinepi.2019.12.015. Epub 2019 Dec 19. PMID 31866471
- [Derived] Burbach JP, Verkooijen HM, Intven M, Kleijnen JP, Bosman ME, Raaymakers BW, van Grevenstein WM, Koopman M, Seravalli E, van Asselen B, Reerink O. RandomizEd controlled trial for pre-operAtive dose-escaLation BOOST in locally advanced rectal cancer (RECTAL BOOST study): study protocol for a randomized controlled trial. Trials. 2015 Feb 22;16:58. doi: 10.1186/s13063-015-0586-4. PMID 25888548
- See also: The PLCRC Project — http://plcrc.nl/